CLINICAL TRIAL: NCT05599503
Title: Social Assistive Robot Interface for People With Alzheimers and Other Dementias to Aid in Care Management
Brief Title: SimpleC Wellness Platform With Social Robot Interaction (Long-term)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SimpleC, LLC (Industry)
Collaborators: University of Georgia (Other); Advanced Medical Electronics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7645D
Record Dates: First submitted 2022-08-30; First posted 2022-10-31 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Engagement, Patient; Quality of Life; Mood; Aging Well; Cognitive Change; Mild Cognitive Impairment; Cognitive Impairment; Dementia
Keywords: At risk, diagnosis
MeSH Terms: conditions — Patient Participation; Cognitive Dysfunction; Dementia; Disease | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SimpleC Wellness Platform with Social Robot Interaction (Experimental): Participants in the Social Robot condition will have access to personal media, reminders, televisit, messaging, news, and wellness programs in their own room via the Companion. Participants will also will have access to social and health reminders as well as social and wellness programs facilitated by a virtual robot agent in their own room via the Companion, social and health reminders as well as social and wellness programs facilitated by a physical robot in the community area and a staff member (likely the activity director).
  Interventions: Behavioral: Behavioral Interventions; Behavioral: Robot Interventions
- SimpleC Wellness Platform (Active Comparator): Participants in the SimpleC Wellness Platform condition will have access to personal media, reminders, televisit, messaging, news, and wellness programs in their own room via the Companion.
  Interventions: Behavioral: Behavioral Interventions

INTERVENTIONS:
Behavioral: Behavioral Interventions — Traditional SimpleC Wellness
Behavioral: Robot Interventions — Robot interventions
  Arms: SimpleC Wellness Platform with Social Robot Interaction

SUMMARY:
This study will be conducted to test a Socially-Assistive Robot (SAR) system for residents in an Assisted Living environment. The goal of the SAR system is to enhance social engagement and connectedness. The system engages residents via robot-facilitated activities such as trivia and reminder and is integrated with the SimpleC Wellness Platform.

DETAILED DESCRIPTION:
This is a mixed-method study to assess the effectiveness of the SAR system. The study includes behavior/lifestyle intervention that are delivered via a robot and/or tablet. The study intervention is a Social Assistive Robot (SAR) System. The SAR system contains the SimpleC Platform, physical robot, virtual agent/robot.

The goal is to engage residents in a natural language conversation as psychosocial support (enhancing mood, mitigating the effects of loneliness, and enhancing social connection and communication) and provide value to the organization and its staff.

Research questions include:

1. Are existing and new residents engaged and satisfied with the Technology Intervention Program?
2. What are the benefits (health, behavioral, economic, and social) of the virtual agent and physical robot?
3. Which users will adopt the SAR system?
4. What are facilitators and barriers to SAR system adoption?
5. Does Technology Acceptance Theory explain adoption over time?
6. Do changing needs affect changing technology attitude?
7. What are guidelines for implementation and design?

Sample: 270 individuals will participate: 90 residents, 90 family, and 90 staff across different study locations. Enrollment will be stopped upon reaching saturation.

1. Participants in both conditions will have access to personal media, reminders, televisit, messaging, news, and wellness programs in their own room via the Companion.
2. Participants in the SAR condition will have access to social and health reminders as well as social and wellness programs facilitated by a virtual robot agent in their own room via the Companion.
3. Participants in the SAR condition will also have access to social and health reminders as well as social and wellness programs facilitated by a physical robot in the community area and a staff member (likely the activity director).

The goal is to offer SAR-facilitated group session at least once per week, for residents to attend at least one such session over the course of the study and two sessions/month.

ELIGIBILITY:
Resident Inclusion Criteria:

* Aged 50+ years
* Any gender
* Fluent in English
* New or current user of SimpleC
* At risk for MCI; MCI; moderate / cognitive impairment (MMSE score of 13 or higher)

Family Member Inclusion Criteria:

* Aged 18+ years
* Any gender
* Fluent in English
* Family or friend of resident
* New or current user of SimpleC
* No diagnosis of dementia or related disorder

Staff Inclusion Criteria:

* Aged 18+ years
* Any gender
* Fluent in English
* Works for the Senior Housing Community
* New or current user of SimpleC

Resident Exclusion Criteria:

* Comorbidities or psychiatric history that would preclude study participation
* Expecting to move during the study (i.e., move out of facility)
* Both legally deaf and blind
* Not able to press tablet buttons
* Not able to verbally answer questionnaires
* Pregnant

Family Caregiver Exclusion Criteria:

* Comorbidities or psychiatric history that would preclude study participation
* Expecting to move during the study (i.e., move out of facility)
* Both legally deaf and blind
* Not able to press tablet buttons
* Pregnant

Staff Exclusion Criteria:

* Expecting to move during the study (i.e., move out of facility)
* Both legally deaf and blind
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Change in Robotic Social Attributes Scale (RoSAS). An 18-item scale with high scores indicating positive attitudes for dimensions of warmth and competency and a negative attitude for dimension of discomfort. | Midpoint (3 months), Final (6 months)
  [Questionnaire] Perception and judgment of Social Assistive Robot social attributes on 3 dimensions: Warmth, competency, and discomfort
Change in Caregiver Guilt Scale. A 4-point scale with higher score indicating higher guilt. | Baseline, Midpoint (3 months), Final (6 months)
  [Questionnaire] Family caregiver feelings of guilt.
Change in Perceived Stress Scale. A 5-point scale with higher scores indicating higher stress. | Baseline, Midpoint (3 months), Final (6 months)
  [Questionnaire] Family caregiver experience of stress in the past 4 months. Modification: Answer as it relates to caregiving.
Change in Technology Acceptance and Experience Questionnaire. A scale with high scores indicating higher acceptance. | Midpoint (3 months), Final (6 months)
  [Questionnaire] Assessment of users' perceived ease of use, usefulness, and satisfaction of using the technology.
Change in Quality of Life. A 13-item survey with high scores indicating higher quality of life. | Baseline, Midpoint (3 months), Final (6 months)
  [Questionnaire] Assessment of different aspects of quality of life, including physical health, energy, family, money.

SECONDARY OUTCOMES:
Technology acceptance and adoption Interview. | Midpoint (3 months)
  [Interview] Assessment of users acceptance and adoption ease of use, usefulness, and satisfaction of using the technology.
Technology acceptance and adoption Interview. | Final (6 months)
  [Interview] Assessment of users acceptance and adoption ease of use, usefulness, and satisfaction of using the technology.
Usability and usefulness | 6 months
  Identified factors that indicate the ease of use and usefulness for different tasks as derived from analysis of: [Interview, usage data]
Conversation quality | 6 months
  [Interview] User perceptions on the usefulness and ease of use in conversing with the technology.
Value proposition/Economic Impact | 6 months
  [Interview] Discussions with facility staff and key decision makers to understand the value of the technology in providing social interaction and reminders to their residents.
Requirements | 6 months
  Identified requirements for design, training, and communication as derived from analysis of: [Interview, observations]
Affect | 6 months
  [Interview] Feelings of enjoyment, satisfaction, when using the technology
Participation Pattern | 6 months
  How often system is used, buttons clicked, voice activation [usage data, interview, observations]

CONTACTS AND LOCATIONS:
Overall Officials: Anne Adams, PhD, Principal Investigator — SimpleC, LLC; Jenay M Beer, PhD, Principal Investigator — University of Georgia
Locations (2):
- United States (2):
  - University of Georgia, Athens, Georgia
  - SimpleC, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No